CLINICAL TRIAL: NCT03825263
Title: Intermittent Pneumatic Compression for Treating Lower Limb Lymphoedema: a Feasibility Study
Brief Title: Intermittent Pneumatic Compression for Treating Lower Limb Lymphoedema
Acronym: IMPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Wales (Other)
Collaborators: Cwm Taf University Health Board (NHS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPRESS
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Lymphoedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Observational control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants receive normal treatment
- Intervention (Experimental): Participants administer Intermittent Pressure Compression using the Lymphassist in addition to normal treatment
  Interventions: Device: Intermittent Pressure Compression

INTERVENTIONS:
Device: Intermittent Pressure Compression — The intervention group use the IPC device for 6 months. Clinic assessment were completed at the beginning and at 3 and 6 months. Participants in the intervention group were invited to use the IPC device twice a day every day during this period.
  Other Names: Lymphassist
  Arms: Intervention

SUMMARY:
The treatment of lymphoedema and its associated complications represent a considerable drain on increasingly limited NHS resources. Intermittent pneumatic compression, specifically the LymphAssist (Huntleigh Healthcare), represents an innovative treatment for this condition but the efficacy of this device needs to be investigated via robust clinical research.

DETAILED DESCRIPTION:
This feasibility study aims to evaluate a proposed methodology designed to assess the efficacy of IPC in the treatment of lymphoedema. The study methodology consisted of a pilot randomised control trial of IPC plus standard lymphoedema care versus standard lymphoedema care alone. Feasibility outcomes included impact on lower limb volume.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over,
* Able to provide written consent,
* Confirmed diagnosis of lower limb ISL stage II or III.

Exclusion Criteria:

Any of these conditions

* Severe congestive heart failure
* Severe skin problems, lower limb ulcers or wounds.
* Presence of cognitive impairment (permanent or intermittent) which would prevent patients from using the IPC device safely or adhering to instructions/study protocol.
* Non-pitting chronic lymphoedema.
* Known or suspected deep vein thrombosis.
* Pulmonary embolism.
* Thrombophlebitis.
* Acute inflammation of the skin (erysipelas, cellulitis).
* Uncontrolled/severe cardiac failure.
* Pulmonary oedema.
* Ischaemic vascular disease.
* Active cancer diagnosis.
* Active metastatic diseases affecting the oedematous region.
* Oedema at the root of the extremity or truncal oedema.
* Severe peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Lower Limb Volume | 3 and 6 months of treatment
  Change in limb volume

SECONDARY OUTCOMES:
Assessment of IPC use on the Quality of Life: QOL Scores | 3 and 6 months
  Change in QOL Scores. Using the Quality of LifeEnjoyment and Satisfication Questionairre short form (Q-LES-Q-SF) with 14 items. Score range is from 14 to 70.
Use of Perometer | 6 months
  Comparison of limb volume measurement methods

CONTACTS AND LOCATIONS:
Overall Officials: Mark Williams, Phd, Principal Investigator — University of South Wales
Locations (1):
- Dewi Sant Hospital, Pontypridd, RCT, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunn N, Williams EM, Fishbourne M, Dolan G, Davies JH. Home management of lower limb lymphoedema with an intermittent pneumatic compression device: a feasibility study. Pilot Feasibility Stud. 2019 Sep 30;5:113. doi: 10.1186/s40814-019-0496-4. eCollection 2019. PMID 31583112